CLINICAL TRIAL: NCT01655589
Title: VEGF Gene Polymorphism and Response to Intravitreal Anti-VEGF Agents in Neovascular Age-related Macular Degeneration
Brief Title: VEGF Gene Association With Response to Neovascular Age-related Macular Degeneration With Anti-VEGF Agents
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institute of Vision, Brasil (Other)
Responsible Party: Sponsor
Other Study IDs: IV-01
Record Dates: First submitted 2012-07-31; First posted 2012-08-02 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-07

CONDITIONS: Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
The main purpose of this study is to investigate the association between VEGF gene polymorphism and the response to intravitreal drugs in neovascular age-related macular degeneration. This is a retrospective review of patients treated between 2008 and 2012 at the Institute of Vision, in Belo Horizonte, Brazil.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of neovascular age-related macular degeneration
* Visual acuity better than 20/400
* Loading dose with three intravitreal injections of anti-VEGF agents, administred one per month over three months
* Follow-up period of at least six months

Exclusion Criteria:

* Choroidal neovascularization secondary to any other cause than age-related macular degeneration
* Eyes with polypoidal choroidal vasculopathy
* Eyes previously submitted to posterior vitrectomy
* Other diseases that could affect visual acuity

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eye clinic in Belo Horizonte, Brazil
Sampling Method: Non-Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2008-01

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Vision, Belo Horizonte, Minas Gerais, Brazil